CLINICAL TRIAL: NCT02973594
Title: Pulse Reduction On Beta-blocker and Ivabradine Therapy
Acronym: PROBE-IT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Heart Association (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 16-1363
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Dilated Cardiomyopathies, Idiopathic; Heart Failure, Systolic; Ventricular Remodeling; Electrical Remodeling
Keywords: left ventricular reverse remodeling; beta-1 adrenergic receptor signaling; idiopathic dilated cardiomyopathy; HCN4 inhibition; beta-1 adrenergic receptor blocker; gene expression
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure, Systolic; Ventricular Remodeling; Atrial Remodeling | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivabradine (Active Comparator): Patients will receive ivabradine 2.5-7.5 mg PO bid in addition to baseline maximum-tolerated beta-blocker therapy.
  Interventions: Drug: Ivabradine
- Placebo (Placebo Comparator): Patients will receive placebo bid in addition to baseline maximum-tolerated beta-blocker therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine
  Other Names: Corlanor
  Arms: Ivabradine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Heart failure with reduced left ventricular ejection fraction (HFrEF) is the most common form of chronic heart failure in subjects ≤ 75 years of age. Beta-blocker therapy greatly reduces mortality and improves ventricular function in HFrEF patients, but 30-40% of patients do not show improvement in ventricular function with beta blockade.

An extensive gene signaling network downstream from the beta1-adrenergic receptor, the primary target of beta-blocker therapy is likely important for development and progression HFrEF. Pathologic changes in this gene signaling network are only reversed towards normal levels when ventricular function improves. One potential mechanism for failure to improve ventricular function in HFrEF patients unresponsive to beta blocker therapy is a lack of heart rate reduction.

Ivabradine is an FDA-approved medication believed to have therapeutic benefit in HFrEF patients through reduction in heart rate independent of beta-blockade. Ivabradine has been shown to reduce the risk of hospitalization for worsening HF in patients with stable, symptomatic chronic heart failure with reduced EF (≤ 35%)in sinus rhythm with resting heart rate ≥ 70 bpm and who are on maximally tolerated doses of beta blockers or who have a contraindication to beta blockers.

Given the high rate of mortality and hospitalization of HFrEF patients even with current therapies, there is a large unmet need for improving HFrEF therapy. The goals of this study are to test the hypothesis that heart rate reduction is an important antecedent for improvement in ventricular function, and to identify components of the beta1-adrenergic receptor gene signaling network responsible for improvement in ventricular function caused by heart rate reduction.

DETAILED DESCRIPTION:
The Pulse Reduction on Beta-blocker and Ivabradine Therapy (PROBE-IT) Study is a double-blind, randomized, two-arm parallel group, placebo-controlled design that compares the effect of heart rate reduction on ventricular reverse remodeling (assessed by LVEF change at 24 weeks) and on the beta1-gene signaling network in NYHA Class I-III HFrEF patients with an idiopathic dilated cardiomyopathy etiology (HFrEF/IDC), who are in sinus rhythm and whose heart rates remain ≥ 70 bpm on target or maximally tolerated doses of beta-blockers to which they have evidence of non-response by LVEF (< 5 absolute percentage points).

Eligible patients will be randomized (2:1) to blinded treatment with ivabradine or matching placebo and will be initiated as per Corlanor® prescribing information over 4 weeks. The dose at 4 weeks post randomization will be considered the intention-to-treat end of titration dose, but further dose adjustment can be made based on clinical factors.

The primary endpoint, i.e., effect of heart rate reduction on reverse remodeling (LVEF), will be assessed after 24 weeks. LV phenotyping by 3D-echocardiography, endomyocardial biopsy and coronary sinus sampling for cardiac norepinephrine levels will be performed at baseline and at 24 weeks. Exercise testing at baseline will be performed to assess level of beta blockade. Upon completion of the study, gene expression in endomyocardial biopsy tissue samples for each patient will be quantified using RNA-seq and quantified with respect to phenotypic measurements including LVEF and heart rate changes.

After the Week 24 Visit, patients will return for an End-of-Study Visit and be offered open label ivabradine with dose initiation accomplished by stopping study drug and starting Corlanor at 5 mg BID or 2.5 mg BID if the patient is taking that dose of study drug. Investigators and patients will not be informed of the blinded study drug assignment at the time of study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. History of non-ischemic (confirmed by coronary angiogram), non-valvular dilated cardiomyopathy considered to be idiopathic, HFrEF NYHA Class I, II, or III.
3. Must have experienced a sign or symptom of clinical heart failure at some time within the preceding 12 months.
4. In sinus rhythm at Screening Visit.
5. Resting HR ≥ 70 bpm at the Screening Visit.
6. Receiving guideline-indicated oral renin-angiotensin-adosterone system (RAAS) inhibitor therapy at the Randomization Visit, i.e., an ACE inhibitor, angiotensin receptor blocker, or sacubitril/valsartan plus a mineralocorticoid receptor antagonist as tolerated.
7. May have ICD or CRT device as indicated.
8. Receiving beta-blocker therapy for ≥ 6 months and target doses for ≥ 3 months prior to Baseline Visit.

   Target dose of carvedilol is 25 mg BID, and metoprolol succinate, 150 mg/day. Patients who are not receiving doses that are at least at these target levels will have their heart failure beta-blocker up-titrated to target and an LVEF re-measured in 3 months, at which time they could be eligible for enrollment. Patients on < target doses who are intolerant to higher than target doses may be enrolled.
9. Evidence of stable or declining LVEF, defined as no increase by ≥ 5 % on a measurement done within 6 months of screening compared to the most recent historical measurement performed within 36 months of the index measure. Must have been on a dose of ≥ 50% of target during the period that documented the lack of a reverse remodeling response. Prior LVEF measurements could have been performed by any imaging technique, e.g., echocardiography, radionuclide methods, MRI, or contrast ventriculography.
10. Women of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at the Baseline and Randomization Visits.

    a. Women who are surgically sterile or post-menopausal for at least 12 months are not considered to be of childbearing potential.
11. Women of childbearing potential must agree to use a highly effective contraception for the duration of the trial and for at least 30 days following the last dose of study drug.
12. Must be competent to understand the information given in the Institutional Review Board (IRB) informed consent form (ICF).
13. Echocardiographic parasternal window adequate for measuring LV volumes by 3D-echo.
14. Must sign the ICF prior to the initiation of any study procedure and not withdraw consent prior to the Randomization Visit.

Exclusion Criteria:

1. NYHA Class IV symptoms at the Randomization Visit.
2. History of HF due to or associated with uncorrected primary valvular disease or history of ischemic heart disease.
3. Any history of atrial fibrillation (even if in sinus rhythm at present).
4. Systolic blood pressure < 90/50 mmHg at the Screening Visit.
5. Significant fluid overload at the Randomization Visit, in the opinion of the Investigator.

   Evidence of significant fluid overload may include:
   1. Mean jugular venous pressure above the clavicle at 90°.
   2. Liver congestion.
   3. Moist pulmonary rales post-cough.
   4. Peripheral edema beyond 1+ pedal not explained by local factors.
6. History of untreated symptomatic bradycardia or if symptomatic bradycardia is likely on full dose of study drug in the opinion of the Investigator.
7. Moderate to severe asthma or other obstructive lung disease requiring chronic use (> 2 days/week) of an inhaled β2-selective adrenergic agonist < 7 days of the Randomization Visit.
8. Untreated thyroid disease, in the opinion of the Investigator, at the Randomization Visit.
9. Serum potassium < 3.5 mmol/L at the Screening Visit.

   a. Lab value will be assessed by the central lab at the Screening Visit and any exclusionary results must be corrected prior to randomization as documented by either the central or local lab.
10. Renal failure requiring dialysis, serum creatinine > 2.5 mg/dL, or an estimated creatinine clearance < 30 mL/min (Cockcroft-Gault) at the Screening Visit.

    a. Lab values will be assessed by the central lab at the Screening Visit and any exclusionary results must be corrected prior to randomization as documented by either the central or local lab.
11. Significant intrinsic liver disease or a total bilirubin > 2.5 mg/dL at the Screening Visit.

    a. Lab value will be assessed by the central lab at the Screening Visit and any exclusionary results must be corrected prior to randomization as documented by either the central or local lab.
12. Participation in a clinical study or treatment with an investigational drug or device within 30 days of the Screening Visit (or 5 half-lives of the investigational agent, whichever is longer).
13. Comorbid condition or illness which, in the opinion of the Investigator, may limit life expectancy to less than 5 years.
14. Serious or active medical or psychiatric condition which, in the opinion of the Investigator, may interfere with treatment, assessment, or compliance with the protocol.
15. History of alcohol, drug, or chemical abuse that, in the opinion of the Investigator, could impair or limit the patient's full participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Left ventricular reverse remodeling according to heart rate response | 24 weeks
  Improvement in left ventricular ejection fraction (LVEF) of ≥ 5 absolute percentage points in patients above vs. below median HR reduction for all subjects.

SECONDARY OUTCOMES:
Comparison of gene expression abundances by heart rate response | 24 weeks
  Quantification of changes in mRNA and microRNA abundance based on response above and below median for all subjects.
Left ventricular reverse remodeling by treatment group (ivabradine vs. placebo) | 24 weeks
  Comparison of change (absolute LVEF percentage points) in subjects randomized to ivabradine vs. placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Bristow, MD PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - The Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of primary data analysis, all gene expression data will be submitted to the Gene Expression Omnibus (GEO). In addition to the standard descriptive and protocol information, the Metadata Spreadsheet will contain subject information required to reproduce primary analyses. Once released by GEO these data will be available for public download. The investigators anticipate this to be complete approximately 2 years after the completion of final subject follow-up.

REFERENCES:
- [Background] Kao DP, Lowes BD, Gilbert EM, Minobe W, Epperson LE, Meyer LK, Ferguson DA, Volkman AK, Zolty R, Borg CD, Quaife RA, Bristow MR. Therapeutic Molecular Phenotype of beta-Blocker-Associated Reverse-Remodeling in Nonischemic Dilated Cardiomyopathy. Circ Cardiovasc Genet. 2015 Apr;8(2):270-83. doi: 10.1161/CIRCGENETICS.114.000767. Epub 2015 Jan 30. PMID 25637602
- [Background] Lowes BD, Zolty R, Minobe WA, Robertson AD, Leach S, Hunter L, Bristow MR. Serial gene expression profiling in the intact human heart. J Heart Lung Transplant. 2006 May;25(5):579-88. doi: 10.1016/j.healun.2006.01.006. Epub 2006 Apr 11. PMID 16678038
- [Background] Lowes BD, Gilbert EM, Abraham WT, Minobe WA, Larrabee P, Ferguson D, Wolfel EE, Lindenfeld J, Tsvetkova T, Robertson AD, Quaife RA, Bristow MR. Myocardial gene expression in dilated cardiomyopathy treated with beta-blocking agents. N Engl J Med. 2002 May 2;346(18):1357-65. doi: 10.1056/NEJMoa012630. PMID 11986409
- [Background] Tardif JC, O'Meara E, Komajda M, Bohm M, Borer JS, Ford I, Tavazzi L, Swedberg K; SHIFT Investigators. Effects of selective heart rate reduction with ivabradine on left ventricular remodelling and function: results from the SHIFT echocardiography substudy. Eur Heart J. 2011 Oct;32(20):2507-15. doi: 10.1093/eurheartj/ehr311. Epub 2011 Aug 29. PMID 21875858
- [Background] Bohm M, Swedberg K, Komajda M, Borer JS, Ford I, Dubost-Brama A, Lerebours G, Tavazzi L; SHIFT Investigators. Heart rate as a risk factor in chronic heart failure (SHIFT): the association between heart rate and outcomes in a randomised placebo-controlled trial. Lancet. 2010 Sep 11;376(9744):886-94. doi: 10.1016/S0140-6736(10)61259-7. PMID 20801495
- [Background] Bristow MR. Treatment of chronic heart failure with beta-adrenergic receptor antagonists: a convergence of receptor pharmacology and clinical cardiology. Circ Res. 2011 Oct 28;109(10):1176-94. doi: 10.1161/CIRCRESAHA.111.245092. PMID 22034480
- [Derived] Altman NL, Gill EA, Kahwash R, Meyer LK, Wagner JA, Karimpour-Fard A, Berning AA, Minobe WA, Carroll IA, Jonas ER, Slavov D, Emani S, Abraham WT, Gollah AR, Ellis SL, Taylor MRG, Graw SL, Mestroni L, McKinsey TA, Buttrick PM, Kao DP, Bristow MR. Heart Rate Reduction Is Associated With Reverse Left Ventricular Remodeling and Mechanism-Specific Molecular Phenotypes in Dilated Cardiomyopathy. Circ Heart Fail. 2025 Apr;18(4):e012484. doi: 10.1161/CIRCHEARTFAILURE.124.012484. Epub 2025 Mar 7. PMID 40052260